CLINICAL TRIAL: NCT06163872
Title: Approaches of Doctors in Different Branches to the Smoking Habits of Their Patients; Patient's Perspective Survey Study
Brief Title: Doctors' Perspective on Tobacco Addiction
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Olcay Ayçiçek, Asist Proff, Karadeniz Technical University
Other Study IDs: Protocol No: 2022/143
Record Dates: First submitted 2023-10-03; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Nicotine Dependence
Keywords: Tobacco; smoking; doctor; patients; health care
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: survey study — survey study

SUMMARY:
ABSTRACT

Aim:

Our study aimed to determine the approaches of our physicians to the smoking habits of their patients other than those with pulmonary diseases.

Method:

Patients examined in different outpatient clinics of our hospital will be asked 7 questions about the doctor's approach to smoking habits.

1) Do you have information about smoking cessation clinic? 2) Has your doctor asked if you smoke? 3) Did he suggest you stop using it? 4) Did he inform you about the relationship between smoking and your disease? 5) Did he provide information about smoking cessation outpatient clinic services? 6) Have you ever thought about quitting smoking after your doctor's briefing? 7) Did you quit smoking after your doctor's briefing?

DETAILED DESCRIPTION:
1. INTRODUCTION:

   Tobacco use can cause many health problems with both its direct effects on all systems and passive smoke exposure (1). Tobacco use is very common in the world and ranks second among the most common causes of death. According to the World Health Organization, 20.2% of people aged 15 and over smoke and more than 8 million people die each year from active smoking. The mortality rates due to passive smoking are too high to be underestimated, and approximately 1.2 million people are lost due to health problems and second-hand smoke exposure (2).

   The prevalence of tobacco use among adults (aged 15 and over) is 31.2% (48% in men and 15% in women). Regular smoking is especially common between the ages of 25-44. Studies show that smoking rates in Turkey are inversely proportional to the level of education (3).

   Physicians are the most influential ones on tobacco use behavior. Informing patients about tobacco addiction, helping with treatment, and drawing a sample profile by not using tobacco is a profile that every physician should portray. Today, smoking cessation support is provided by specialist physicians (Chest diseases, Family medicine) to help smokers quit. In this process, patients are supported with both behavioral treatment and medical treatment (4-5). However, this support should not be limited to the specified sections. The physician evaluating a patient should contribute to tobacco control regardless of his/her branch, learn whether the patient is using tobacco or not, advise the patient to quit if he/she is using it, and should inform and direct the patient from smoking cessation outpatient clinics.

   In this study, it is aimed to evaluate the attitudes and habits of our physicians working in non-chest disease departments in our hospital and to determine their role in developing a positive attitude towards patients. With the results of the study, it is aimed to question the smoking habits of physicians in patients, to be a guide and leader, to reveal the differences in physician approaches according to branches, to be a guide for initiatives to increase positive attitudes by analyzing positive and negative results and self-criticism.
2. MATERIALS-METHODS:

The study will start after the approval of the faculty ethics committee. Patients who were examined in other branch outpatient clinics other than the chest diseases department of our hospital will questioned for 3 months. Those who did not volunteer to participate in the survey, patients under the age of 18, and patients whose mental status was not suitable for the survey will not included in the study. As the place where the questionnaire will be conducted, the blood collection laboratory where all the patients come mostly was chosen, and the patients who came here to donate blood were randomly selected and the questionnaire was conducted. In addition to their demographic characteristics, the following 7 questions were asked to the patients. 1) Do you know about smoking cessation outpatient clinic? 2) Has your doctor asked if you smoke? 3) Has he suggested you stop using it? 4) Has he informed you about the relationship of smoking with your illness? 5) Has s/he informed about smoking cessation outpatient clinic services? 6) Have you ever considered quitting smoking after your doctor's briefings? 7) Have you quitted smoking after your doctor's briefings? The responses will compared according to the branches.

It will investigated whether the patients asked the questions specified in the data form about their demographic characteristics, educational status, diagnosis, the branch they were examined in, the recommendations of the examining physician regarding the patient's smoking habit and whether they quit if they smoked.

2.1.Statistical Analysis The suitability of the data for normal distribution will examined with the ShapiroWilk and Kolmogorog Smirnov tests. Kruskall-Wallis, Mann-Whitney U, student-t and chi-square tests will used for intergroup comparisons. General linner modeling, Wilcowon and Friedman tests will used in serial follow-up data. Data will presented as percentage, mean (std deviation) and median (minimum-maximum). Pearson's chi-square test will used to compare the qualitative data. Categorical data will presented as frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were examined in other branch outpatient clinics other than the chest diseases department of our hospital

Exclusion Criteria:

* Those who did not volunteer to participate in the survey
* Patients under the age of 18
* patients whose mental status was not suitable for the survey

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were examined in other branch outpatient clinics other than the chest diseases department of our hospital
Sampling Method: Non-Probability Sample
Enrollment: 941 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Nicotine addiction | 3 month
  Determining how effective doctors working in branches other than pulmonology are in helping smokers quit smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Ozdogan Algın, MD, Study Chair — Karadeniz Technical University Faculty of Medicine Department of Chest disease; Ensar Cihad Emiroglu, MD, Study Chair — Karadeniz Technical University Faculty of Medicine Department of Chest disease; Funda Oztuna, Proff, Study Chair — Karadeniz Technical University Faculty of Medicine Department of Chest disease
Locations (1):
- Department of Chest Diseases, Division Of Intensive Care Medicine, Faculty of Medicine, Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided